CLINICAL TRIAL: NCT02519426
Title: Clinical Validation of a Novel Classification for Predicting Surgical Complexity of Impacted Mandibular Third Molar Extraction: an Observational Clinical Trial
Brief Title: Clinical Validation of a Novel Classification for Predicting Surgical Complexity in Mandibular Wisdom Teeth Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: University of Trieste (Other)
Responsible Party: Principal Investigator, Povilas Daugela, Assistant, Lithuanian University of Health Sciences
Other Study IDs: J&D Classification Validation
Record Dates: First submitted 2015-08-03; First posted 2015-08-11 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Impacted Third Molar Tooth; Tooth Extraction Status Nos
Keywords: Third molar; Classification; Inferior alveolar nerve; Lingual nerve injuries; Mandibular canal
MeSH Terms: conditions — Lingual Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Cumulative complexity score <9: Mandibular third molar surgery patients with Juodzbalys and Daugela impacted mandibular third molars surgical extraction complexity index cumulative score lower than 9.
  Interventions: Procedure: Mandibular third molar surgery
- Cumulative complexity score y≥9: Mandibular third molar surgery patients with Juodzbalys and Daugela impacted mandibular third molars surgical extraction complexity index cumulative score higher than 9.
  Interventions: Procedure: Mandibular third molar surgery
- Pell Gregory index <Class 2B: Mandibular third molar surgery patients with Pell Gregory index Class 1A, Class 1B, Class 1C, or Class 2A
  Interventions: Procedure: Mandibular third molar surgery
- Pell Gregory index ≥Class 2B: Mandibular third molar surgery patients with Pell Gregory index Class 2B, Class 2C, Class 3A, Class 3B, or Class 3C
  Interventions: Procedure: Mandibular third molar surgery
- Winter index <Horizontal impaction: Mandibular third molar surgery patients with Winter predicted index of Mesio-Angular, Disto-Angular or Vertical impaction
  Interventions: Procedure: Mandibular third molar surgery
- Winter index ≥Horizontal impaction: Mandibular third molar surgery patients with Winter predicted index of Horizontal, Buccal / Lingual Obliquity, Transverse, Inverse impaction
  Interventions: Procedure: Mandibular third molar surgery

INTERVENTIONS:
Procedure: Mandibular third molar surgery — Mandibular third molar surgery is a mandibular wisdom tooth removal procedure in which surgical access is required to completely remove a tooth. Even if the tooth is visible in the mouth without surgically exposing it, surgical techniques may be necessary to remove the tooth. This includes sectioning the tooth into two or more pieces, corticotomy, and removal with forceps and elevators, whether or not a soft tissue incision is made.

SUMMARY:
The study evaluates and validates a new classification proposed by Juodzbalys and Daugela in 2013 predicting the complexity of impacted mandibular third molars surgical extraction, comparing it with other two, scientifically approved (Pell and Gregory, Winter) classifications.

DETAILED DESCRIPTION:
The extraction of mandibular impacted wisdom teeth is the most widespread surgical procedure performed in oral surgery. There are many situations indicating the extraction of those teeth as well as risks and protective factors that may contraindicate it. A reliable classification predicting the complexity of the surgical procedure and the related risk of complications would greatly help the surgeon in the diagnostic phase.

The aim of the study is to evaluate if the classification proposed by Juodzbalys and Daugela in 2013 could be effective in predicting the complexity of impacted mandibular third molars surgical extraction, and to compare its effectiveness with commonly used Pell and Gregory, Winter classifications.

A blind expert surgeon will assess postoperatively all CBCTs (Cone beam computed tomographies) and OPGs (orthopantomographs) not older than 12 months, and will assign the score for each extracted tooth for the three classification (Juodzbalys and Daugela - Pell and Gregory - Winter). Duration of the surgical procedure, assessment of the surgical technique and of intra- and post-operative complications will be considered as the main parameters to evaluate surgical difficulty. VAS (Visual Analogue Scale) pain score and NSAID (Nonsteroidal anti-inflammatory drug) pills count taken by each patient of the 7 days postoperative period will be also evaluated.

Statistical unit analyzed will be the single tooth. It should be noted that if a single patient has a bilateral impacted tooth to be extracted it will be randomly selected only one to be analyzed. Patients will be divided into two groups according to Juodzbalys and Daugela classification score (x<9≤y), two groups according to each predicted extraction difficulty to Pell Gregory (x<Class 2B≤y) and Winter (x<Horizontal impaction≤y) classifications.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with an age comprised between 16 to 90 years
* Healthy patients ( ASA (American Society of Anesthesiologists) Physical status index ≤ 2)
* CBCT and/or OPG performed not before than 12 months before surgery
* Complete roots formation of 38 or 48 at CBCT and/or OPG examination
* Signed informed consent

Exclusion Criteria:

* Smoking > 10 cigarettes per day
* Presence of any neoplastic lesion (benign or malignant), clinically or radiologically evaluable, at the site or close to the impacted tooth
* Presence of any radiolucent lesion >1 cm at impacted tooth level

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total number of 110 (including eventual drop outs) third molar surgery patients will be selected randomly. One tooth per patient is going to be evaluated. It should be noted that if a single patient has a bilateral impacted tooth to be extracted it will be randomly selected only one to be analyzed. In total 104 extraction are going to be evaluated. Patients will be divided into two groups according to Juodzbalys and Daugela classification score (x<9>y). Sample size of 52 subjects per group was calculated to detect a mean difference between the two groups of 10 minutes with an expected SD of 18 minutes. Power was set at 80% and alpha at 0.05.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Duration of the mandibular third molar surgery | Up to 2 hours
  Duration of the surgical procedure is counted from the beginning of surgical manipulations to complete removal of mandibular wisdom tooth and wound closure if applicable.

SECONDARY OUTCOMES:
Composite assessment of the surgical technique and of intra - and post-operative complications | 7 days
  Surgical approach (open flap, flapless), surgical technique (simple mobilization of the tooth, ostectomy, coronectomy, roots separation), used surgical devices (forceps and elevators, rotary carbide bur, rotary diamond bur, piezosurgery), as well as intra-operative side effects (apex fracture, inferior alveolar artery bleeding, fragment displacement in soft tissues, mandible fracture) and type of wound are evaluated.
Pain and Discomfort assessment with VAS scale | 7 days
  surgery with 10 grade VAS scale, where 0=no pain, 10=Worst possible, unbearable, excruciating pain.
NSAID assumption | 7 days
  Patient every day NSAID (Ibuprofen 400 mg) tablet count taken in in the consecutive 7 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, DDS,MSc,Prof, Study Chair — The University of Trieste; Gintaras Juodzbalys, DDS,PhD,Prof, Study Chair — The Lithuanian University of Health Sciences; Povilas Daugela, DDS, Assist., Principal Investigator — The Lithuanian University of Health Sciences; Federico Berton, DDS, Principal Investigator — The University of Trieste; Teresa Lombardi, DDS, Principal Investigator — The University of Trieste; Roberto Di Lenarda, DDS,MSc,Prof, Principal Investigator — The University of Trieste; Tautvydas Andriulionios, DDS, Principal Investigator — The Lithuanian University of Health Sciences
Locations (2):
- The University of Trieste, Trieste, Italy
- Lithuanian University of Health Sciences, Kaunas, Lithuania

REFERENCES:
- [Background] Juodzbalys G, Daugela P. Mandibular third molar impaction: review of literature and a proposal of a classification. J Oral Maxillofac Res. 2013 Jul 1;4(2):e1. doi: 10.5037/jomr.2013.4201. PMID 24422029